CLINICAL TRIAL: NCT05655962
Title: A Structured Framework for Assessment of Rehabilitation and Sicklisting (STARS) in Primary Care - Evaluating Effects, Professionals' and Patient Experiences of STARS
Brief Title: A Structured Framework for Assessment of Rehabilitation and Sicklisting in Primary Care - a Multicenter Study
Acronym: STARS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Östergötland (Other)
Collaborators: Region Jönköping County (Other Government); Kalmar County Hospital (Other)
Responsible Party: Principal Investigator, Hanna Israelsson Larsen, PhD, MD, Adjunct senior lecturer, Region Östergötland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-04412
Record Dates: First submitted 2022-11-30; First posted 2022-12-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Public Health

STUDY DESIGN:
Intervention Model Description: 9 centers implement the STARS framwork, and are compared to control centers that do not work according to STARS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STARS center (Experimental): Centers in the southeast region of Sweden working according to STARS.
  Interventions: Other: STARS
- Control center (No Intervention): Centers in the southeast region of Sweden not working according to STARS.

INTERVENTIONS:
Other: STARS — STARS is a structured framework for assessment of rehabilitation and sicklisting, applied by primarily the rehabilitation coordinators working at the primary health care centers.
  Arms: STARS center

SUMMARY:
In a controlled pragmatic multicenter primary care study, centers working according to a newly constructed structured framework for assessment of rehabilitation and sicklisting (STARS) will be investigated. Nine intervention centers working according to STARS will be compared to matched control centers not working according to STARS. The design of this study includes qualitative as well as quantitative measures, with the aim to evaluate the effects of STARS at patient, staff, and organization levels.

DETAILED DESCRIPTION:
Common mental disorders and musculoskeletal pain are the most frequent causes for sick leave. Despite frequent appearance, the sick listing process is often perceived as uncertain and unclear, both among sick listed patients and health care professionals. In addition, the follow-up of patients on sick leave is sometimes lacking, leading to protracted processes and suffering for the patients. In three healthcare regions in the Southeast of Sweden, a structured framework regarding the sick listing and rehabilitation process has been developed in close collaboration between researchers and clinicians: STructured Assessment of Rehabilitation and Sick listing in primary care (henceforth referred to as STARS), to meet the needs among patients and professionals within health care, as well as to meet the statutory demands regarding coordination efforts for sick-listed patients. The comprehensive design of this study includes qualitative as well as quantitative studies, with the aim to evaluate the effects of STARS at patient, staff, and organization levels.

In a controlled pragmatic multicenter primary care study, nine centers (three from each region) working according to STARS will be compared with control centers with care as usual. The STARS framework has seven detailed method supports for health care professionals, each to be applied at different times during the first 90 days of the patients´ sick listing. Potential study participants are a) patients aged 18-65 that are sick listed due to common mental disorders, musculoskeletal pain or residual symptoms from Covid-19 and; b) medical staff involved in the sick listing- and rehabilitation process. Data will be collected through focus group interviews (health care professionals), individual interviews (patients), questionnaires (patients and health care professionals) as well as national registries regarding length and extent of sick listing. Primary outcome measures are length and extent of sick listing up until 90 days (quantitative) and the medical staffs´ experiences and perceptions regarding following the guidelines of the STARS framework (i.e. both qualitative and quantitative data). Secondary outcome measures at the included STARS centers are i) the patients' experiences regarding their sick listing process, ii) the medical staffs´ experiences of their organizational work environment , iii) causes for sick listing >90 days, and iv) health economic studies to investigate the cost-effectiveness of STARS.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* age ≥18 years;
* sick-listed due to ICD-diagnoses: F00-F99 (mental/behavioral disorders), M00-99 (musculoskeletal pain), R52 (non-specified pain), U08.9, U09.9 or U10.9 (codes related to COVID19);
* have received rehabilitation coordination performed by a RECO

Health care professionals:

- Health care professionals involved in the sick-listing process of the patients at the health care center.

Exclusion Criteria:

Patients:

* inability to understand Swedish;
* incapacity to give informed consent;
* protected identity

Health care professionals:

- Health care professionals not involved in the sick-listing process of the patients at the health care center.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative measures regarding the patients' perception of STARS, assessed by interviews. | Through study completion, an average of 2 years.
  The patients' perceptions and experiences of their sick listing process at STARS centers, as described in individual interviews with the study participants.
Length of sick leave in days. | Through study completion, an average of 2 years.
  Number of days on the sick leave for patients receiving care at a STARS center compared to control centers.

SECONDARY OUTCOMES:
Qualitative measures regarding the healthcare professionals' perception of STARS, assessed by interviews. | Through study completion, an average of 2 years.
  The health care professionals' perceptions and experiences of the sick listingprocess at STARS centers.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna I Larsen, Principal Investigator — Region Östergötland
Locations (1):
- Region Östergötland, Norrköping, Sweden

IPD SHARING:
Plan to Share IPD: No